CLINICAL TRIAL: NCT05202067
Title: Impact of Pharmaceutical Education on Medication Adherence in Patients With Type 2 Diabetes Mellitus and Systemic Arterial Hypertension Treated at the Hospital Civil de Guadalajara "Dr. Juan I. Menchaca"
Brief Title: Impact of Pharmaceutical Education on Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Civil Juan I. Menchaca (Other)
Collaborators: Drake University (Other)
Responsible Party: Principal Investigator, Abelardo Contreras Vergara, Principal Investigator, Hospital Civil Juan I. Menchaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0269/18/HCJIM/01
Record Dates: First submitted 2021-12-22; First posted 2022-01-21 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes; Systemic Arterial Hypertension; Medication Adherence
Keywords: Pharmaceutical education; Type 2 Diabetes Mellitus; Systemic Arterial Hypertension; Medication adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Medication Adherence

STUDY DESIGN:
Intervention Model Description: The patients assigned to the intervention group will receive from the research pharmacist, a didactic talk (of at least 10 and up to 20 minutes), where they will be provided information about type 2 diabetes mellitus and Systemic Arterial Hypertension, causes of the disease and consequences of poor control, on its pharmacological treatments, changes in lifestyle and diet. In addition, the patient will be given an updated list of their prescribed medications on a wallet card.
  Patients assigned to the control group will receive only standard care, represented by regular consultation with their prescribing physician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pharmaceutical education (Experimental): The patients assigned to the intervention group will receive from the research pharmacist, a didactic talk (of at least 10 and up to 20 minutes), where they will be provided information about type 2 diabetes mellitus and Systemic Arterial Hypertension, causes of the disease and consequences of poor control, on its pharmacological treatments, changes in lifestyle and diet. In addition, the patient will be given an updated list of their prescribed medications on a wallet card.
  Interventions: Behavioral: pharmaceutical education
- control (No Intervention): Patients assigned to the control group will receive only standard care, represented by regular consultation with their prescribing physician.

INTERVENTIONS:
Behavioral: pharmaceutical education — The patients who were assigned to the intervention group will receive a didactic talk from the research pharmacist. In addition, the patient will be given an updated list of their prescribed medications on a wallet card.
  Arms: pharmaceutical education

SUMMARY:
Purpose. To evaluate the impact of pharmaceutical education in patients with Type 2 Diabetes Mellitus and Systemic Arterial Hypertension on their medication adherence.

Material and research methods. Randomized clinical trial with a control group with a duration of 6 months of follow-up. Patients with a diagnosis of Type 2 Diabetes Mellitus andWE Systemic Arterial Hypertension treated in the internal medicine outpatient of a school hospital will be included. Adherence to medication will be evaluated using Morisky's 8-item medication adherence scale.

The investigators believe that Pharmaceutical education increases therapeutic adherence in patients with Type 2 Diabetes Mellitus and Systemic Arterial Hypertension.

DETAILED DESCRIPTION:
Patients and study design In this randomized and controlled clinical trial, patients will be assigned to two study groups: intervention group and control group; The patients will be followed for 6 months, considering evaluations at 0, 3 and 6 months.

To improve patient adherence to treatment, the investigators will provide a pocket card with an up-to-date list of the patient's prescribed medications along with recommendations for follow-up care. For the evaluation of adherence to treatment, © MMAS is used, it is authorized: MMAR, LLC., Donald E. Morisky # 6533-7069-1342-3041-5361, 294 Lindura Court, Las Vegas, Nevada 89138-4632.

Variables analyzed After randomization, the investigator will interview patients to obtain demographic data and their medical history. Data such as: time of evolution of the disease, number of prescribed medications, family support, cost of drug treatments will be collected, and the levels of glycosylated hemoglobin, fasting plasma glucose, cholesterol and triglycerides will be determined.

Medication adherence Adherence to medication will be evaluated using the Morisky method of 8 items, which is a validated indicator of non-compliance with medication in the treatment of chronic diseases, the Morisky Medication Adherence Scale It is a generic scale to evaluate the patient's behavior regarding adherence to treatment, the points obtained with MMAS-8 are added to give a range of low, medium and high adherence scores. The total score is a sum of the 8 items and ranges between 0 and 8: values with a score greater than 8 reflect high adherence to medication, values between 6 and 7 reflect medium adherence and values below 6 reflect low adherence.

Sample size calculation A sample size calculation shows that a sample of 38 patients in each group is sufficient to find a difference in adherence to treatment with an alpha error of 0.05 and a power of 0.80 of the test, contemplating a 20% loss. The calculation was performed with the expected proportions formula.

Statistical analysis The investigators will report categorical variables as frequencies and percentages and analyzed with χ2 or Fisher's exact tests as necessary; quantitative variables will be presented as mean and standard deviation. The investigators will use the Wilcoxon test for intragroup comparisons and the Mann-Whitney U test for intergroup comparisons. The results will be considered significant at a two-sided p value of <0.05, with a 95% confidence interval. The statistical analyzes will be carried out using Statistical Solutions for Products and Services version 24.0.

ELIGIBILITY:
Inclusion Criteria:

* Patients cared for by the internal medicine outpatient area of the OPD Nuevo Hospital Civil de Guadalajara "Dr. Juan I. Menchaca "
* 18-60 years
* Both genres
* With a diagnosis of type 2 diabetes mellitus and systemic arterial hypertension
* That they gave their consent under information

Exclusion Criteria:

* Inpatients on the day of their internal medicine outpatient appointment.
* Patients for whom pharmacological treatment was not prescribed for the treatment of DM2 and SAH.
* Patients who do not speak Spanish.
* Patients who could not or could not read.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Medication adherence | Basal
  Adherence to medication will be evaluated using the Morisky method of 8 items, which is a valid indicator of non-compliance with medication in the treatment of chronic diseases, the Morisky Medication Adherence Scale is a generic scale to evaluate the behavior of the patient regarding adherence to treatment, the articles obtained with MMAS-8 are added to give a range of low, medium and high adherence scores.
Medication adherence | 3 months
  Adherence to medication will be evaluated using the Morisky method of 8 items, which is a valid indicator of non-compliance with medication in the treatment of chronic diseases, the Morisky Medication Adherence Scale is a generic scale to evaluate the behavior of the patient regarding adherence to treatment, the articles obtained with MMAS-8 are added to give a range of low, medium and high adherence scores.
Medication adherence | 6 months
  Adherence to medication will be evaluated using the Morisky method of 8 items, which is a valid indicator of non-compliance with medication in the treatment of chronic diseases, the Morisky Medication Adherence Scale is a generic scale to evaluate the behavior of the patient regarding adherence to treatment, the articles obtained with MMAS-8 are added to give a range of low, medium and high adherence scores.

CONTACTS AND LOCATIONS:
Overall Officials: SELENE v HUERTA, PhD, Principal Investigator — Universidad De Guadalajara (UDG)
Locations (1):
- Hospital civil de Guadalajara "Dr. Juan I. Menchaca", Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793